CLINICAL TRIAL: NCT03055780
Title: Clinical Trial for SURECardio CT-FFR
Brief Title: Diagnostic Accuracy to Detect Hemodynamically Significant Stenosis by Non-invasive SURECardio CT-FFR
Status: Completed | Type: Observational
Sponsor: Toshiba Medical Systems Corporation, Japan (Industry)
Responsible Party: Sponsor
Other Study IDs: SGD03-0667
Record Dates: First submitted 2017-02-14; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- CT-FFR. CTA. FFR: 59 patients with suspected CAD that have been scheduled for an interventional FFR study
  Interventions: Device: CT-FFR. CTA. FFR

INTERVENTIONS:
Device: CT-FFR. CTA. FFR — Study is to compare results of CT FFR against CTA and interventional FFR

SUMMARY:
The aim of this study was to determine the diagnostic accuracy of SURECardio CT-FFR to detect functionally significant coronary stenosis.

DETAILED DESCRIPTION:
CT acquision and invasive FFR measurement is performed for each patients. The diagnostic accuracy of coronary CTA and SURECardio CT-FFR is investigated using Invasive FFR is used as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* suspected coronary artery disease
* hemodynamically stable condition

Exclusion Criteria:

* hemodynamic instability
* atrial fibrillation
* morbid obesity (BMI≥40 kg/m2)
* previous stent implantation
* recent myocardial infarction (within 30 days)
* age <40 years
* renal insufficiency (eGFR <60mL/min/1.73m2)
* bronchospastic lung disease requiring long term steroid therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected coronary artery disease
Sampling Method: Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of SURECardio CT-FFR to detect functionally significant coronary stenosis | one day

IPD SHARING:
Plan to Share IPD: No